CLINICAL TRIAL: NCT00063700
Title: Impact of Non-Commercialism Policy in Seattle Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Purpose: Prevention
Other Study IDs: INCPSS (completed)
Record Dates: First submitted 2003-07-02; First posted 2003-07-03 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Obesity
Keywords: obesity in school aged children
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Procedure: reducing exposure to marketing pressures

SUMMARY:
This pilot study on the impact of a non-commercialism policy in Seattle schools will assess and evaluate obesity-related health outcomes of a real-life policy decision, recently voted on and adopted by the Seattle School Board. The policy reduces the exposure to advertising and other marketing pressures, including those from commercial food vendors.

ELIGIBILITY:
no restrictions

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Dates: Start 2002-09; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle school, Seattle, Washington, United States